CLINICAL TRIAL: NCT01351519
Title: A Phase 2 Study of Aminolevulinic Acid (ALA) to Enhance Visualization and Resection of Malignant Glial Tumors of the Brain
Brief Title: A Study of Aminolevulinic Acid Used to Enhance Visualization and Surgical Removal of Brain Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Limited staff available for enrollment and limited availability of drug
Sponsor: MultiCare Health System Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALA 11.07
Record Dates: First submitted 2011-05-07; First posted 2011-05-11 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Malignant Glioma; Glioma; Glioblastoma; Glioblastoma Multiforme; Astrocytoma
Keywords: Glioma; Glioblastoma; Glioblastoma Multiforme; Astrocytoma; Brain Tumor
MeSH Terms: conditions — Glioma; Glioblastoma; Astrocytoma; Brain Neoplasms | interventions — Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aminolevulinic Acid (AL) (Experimental)
  Interventions: Drug: Aminolevulinic Acid

INTERVENTIONS:
Drug: Aminolevulinic Acid — Aminolevulinic Acid will be administered as a single oral dose of 20mg/kg given in 50ml of water three hours before surgery.
  Other Names: ALA; 5-Aminolevulinic Acid; Levulan

SUMMARY:
In this study subjects will be administered a single oral dose of Aminolevulinic Acid (ALA) prior to surgical resection of their brain tumor. The ALA ultimately causes brain tumor tissue to fluoresce or light up under ultraviolet light. During surgery an ultraviolet light in the microscope chain will be turned on. The tumor tissue will fluoresce bright pink allowing the surgeon to more easily differentiate tumor tissue from normal brain tissue. The aim of the study is to determine whether ALA and fluorescent visualization of tumor tissue improves the surgeon's ability to completely resect or remove the brain tumor.

DETAILED DESCRIPTION:
This is a Phase 2 study and all subjects will receive open label Aminolevulinic Acid in a dose of 20mg/kg given orally 3 hours prior to surgery. Brain tumors will be resected with the aid of ultraviolet light to visualize the tumor. After surgery an MRI will be done to determine whether the tumor has been completely or partially resected. All subjects will be followed for safety. All subjects will be followed closely by clinical examination and by MRI to monitor for disease recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Clinically documented primary brain tumor for which surgical resection is indicated.
* Age 18 years and older.
* ECOG Performance status less than or equal to 2.
* Laboratory values as follows:

Leukocytes greater than or equal to 3,000. ANC greater than or equal to 1,500. Platelets greater than or equal to 100,000. Total Bilirubin WNL. AST/ALT less than or equal to 2.5 times ULN. Creatinine WNL. or Creatinine Clearance greater than or equal to 60ml/min/1.73m2 if SCr above institutional normal.

-Ability to provide informed consent or consent from a Legally Authorized Representative.

Exclusion Criteria:

* Receipt of an investigational agent within 30 days.
* Allergy to ALA or similar compounds.
* Personal or family history of porphyria.
* Uncontrolled intercurrent illness.
* Inability to comply with the protocol.
* Pregnancy, breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Time to disease progression after initial surgery. | Up to 2 years
  Determine time-to-progression compared to that in comparable cases performed without the aid of ALA.
Complete Resection | Day 2
  Determine the percentage of patients with complete resections of contrast-enhancing tumor, compared to historical controls

SECONDARY OUTCOMES:
Determine the number of subjects with adverse events due to ALA in this dosage and indication. | Through 45 days
  Subjects will be followed closely for adverse events including biochemical abnormalities through laboratory monitoring and for clinically evident adverse events including possible skin reactions that may occur.
Overall Survival | Up to three years
  Determine the overall survival compared to historical controls.

CONTACTS AND LOCATIONS:
Overall Officials: William Morris, MD, Principal Investigator — MultiCare Health System; Richard Shine, PharmD, BCPS, Study Director — MultiCare Health System Research Institute
Locations (1):
- MultiCare Health System Research Institute, Tacoma, Washington, United States

REFERENCES:
- [Result] Stummer W, Pichlmeier U, Meinel T, Wiestler OD, Zanella F, Reulen HJ; ALA-Glioma Study Group. Fluorescence-guided surgery with 5-aminolevulinic acid for resection of malignant glioma: a randomised controlled multicentre phase III trial. Lancet Oncol. 2006 May;7(5):392-401. doi: 10.1016/S1470-2045(06)70665-9. PMID 16648043